CLINICAL TRIAL: NCT00127179
Title: MK0906 Phase III Double-Blind Comparative Study - Benign Prostate Hyperplasia
Brief Title: A Study of an Investigational Study Drug for Benign Prostatic Hyperplasia (0906-140)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0906-140; MK0906-140; 2005_042
Record Dates: First submitted 2005-08-03; First posted 2005-08-05 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Finasteride; Duration of Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0906, finasteride / Duration of Treatment: 48 weeks
Drug: Comparator: placebo / Duration of Treatment: 48 weeks

SUMMARY:
The purpose of this trial is to determine the efficacy and safety of an investigational drug in patients with benign prostatic hyperplasia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with benign prostatic hyperplasia

Exclusion Criteria:

* Patients who are suspected to be suffering from prostatic cancer

Ages: 50 Years to 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2004-01-01 (Actual); Primary Completion 2005-07-01 (Actual); Study Completion 2005-07-25 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the International Prostate Symptom Score

SECONDARY OUTCOMES:
Change from baseline in QOL - index
Change from baseline in maximum urinary flow rate, %
Change from baseline in Prostate volume

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC